CLINICAL TRIAL: NCT00318227
Title: Evaluation of a Liberal Versus Restrictive Blood Transfusion Strategy in Elderly Patients Following Coronary Bypass or Aortic Valve Surgery
Brief Title: Randomized Trial of a Liberal Versus a Restrictive Transfusion Strategy in Elderly Cardiac Surgery Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R-03-043; 9540
Record Dates: First submitted 2006-04-24; First posted 2006-04-26 (Estimated); Last update posted 2017-08-28 (Actual); Status verified 2017-08

CONDITIONS: Anemia; Coronary Artery Bypass Surgery
Keywords: Postoperative care; Cardiac Surgery; Blood Transfusion
MeSH Terms: conditions — Anemia | interventions — Blood Transfusion

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Liberal Red cell transfusion arm (Active Comparator): Transfusion if Hgb <100g/L
  Interventions: Procedure: Blood Transfusion
- Restrictive Red Cell transfusion (Active Comparator): Transfusion if Hgb <70g/L
  Interventions: Procedure: Blood Transfusion

INTERVENTIONS:
Procedure: Blood Transfusion — Blood transfusion will be administered when the transfusion trigger is met.

SUMMARY:
The purpose of this study is to determine whether a less restrictive strategy of red blood cell transfusion in elderly patients following coronary bypass surgery results in enhanced postoperative recovery as determined by quality of life assessment, exercise tolerance and clinical outcomes.

Two postoperative transfusion strategies:

1. Liberal - transfused when Hgb is <100g/L
2. Restrictive - transfused when Hgb is <70g/L

ELIGIBILITY:
Inclusion Criteria:

* Patients >=70 years of age undergoing non-emergency coronary artery bypass surgery
* Initial postoperative hemoglobin level 70-90g/L

Exclusion Criteria:

* Patients who are unable to provide informed consent in English
* Patients with preoperative hemoglobin concentrations <100g/L
* Patients who require emergency re-operation
* Patients with intraoperative or postoperative bleeding diathesis
* Patients with postoperative clinical instability (eg. low output state)
* Patients in whom insertion of an intra-aortic balloon pump is required

Ages: 70 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 73 (Actual)
Dates: Start 2004-06-21 (Actual); Primary Completion 2009-04-21 (Actual); Study Completion 2010-02-23 (Actual)

PRIMARY OUTCOMES:
Distance walked during 6 minute walk test at 5 weeks postop | 5 weeks

SECONDARY OUTCOMES:
renal failure, hospital length of stay, Quality of Life questionnaire | during hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Mary Lee Myers, MD FRCSC, Principal Investigator — London Health Sciences Centre/University of Western Ontario; Robin Varghese, MD MS FRCSC, Principal Investigator — London Health Sciences Centre/University of Western Ontario
Locations (1):
- London Health Sciences Centre - University Campus, London, Ontario, Canada

REFERENCES:
- [Derived] Carson JL, Stanworth SJ, Dennis JA, Fergusson DA, Pagano MB, Roubinian NH, Turgeon AF, Valentine S, Trivella M, Doree C, Hebert PC. Transfusion thresholds and other strategies for guiding red blood cell transfusion. Cochrane Database Syst Rev. 2025 Oct 20;10(10):CD002042. doi: 10.1002/14651858.CD002042.pub6. PMID 41114449